CLINICAL TRIAL: NCT02333760
Title: Long Term Safety Follow up of Patients Enrolled in the Phase I/II Clinical Trial of Haematopoietic Stem Cell Gene Therapy for the Wiskott Aldrich Syndrome (GTG002-07 and GTG003-08).
Brief Title: Long Term Safety Follow up of Haematopoietic Stem Cell Gene Therapy for the Wiskott Aldrich Syndrome
Acronym: WASFUP
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genethon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GNT-WAS-03
Record Dates: First submitted 2014-10-28; First posted 2015-01-07 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Wiskott-Aldrich Syndrome
MeSH Terms: conditions — Wiskott-Aldrich Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: Autologous CD34+ cells transduced with WASP lentiviral vector — Follow up of ex vivo gene therapy transplantation of patient's autologous CD34+ cells transduced with lentiviral vector containing human WASP gene

SUMMARY:
An open follow up study of patients enrolled in the Phase 1/2 clinical trial of haematopoietic stem cell gene therapy for the Wiskott-Aldrich Syndrome and treated with autologous CD34+ cells transduced with the w1.6_hWASP_WPRE (VSVg) lentiviral vector.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in the initial phase I/II WAS conducted in France and United Kingdom (GTG002.07 and GTG003.08).
* Parents, guardians or patient signed informed consent, guardians or patient signed informed consent

Exclusion Criteria:

• Parents, guardians, patients unwilling to return for the follow up study period.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-09; Primary Completion 2032-10 (Estimated); Study Completion 2032-10 (Estimated)

PRIMARY OUTCOMES:
Incidence and type of SAEs | yearly from 3 years to 15 years
  Incidence and nature of delayed events such as malignancies, hematologic, autoimmune events, mortality
Lentiviral integration sites | yearly from 3 years to 15 years (from 11 to 15 yearly time points, only in case of Advers Events of Special Interest)
  Presence of lentiviral integration sites in different cells sub-populations
Vector copy numbers | yearly from 3 years to 15 years (from 11 to 15 yearly time points, only in case of Advers Events of Special Interest)
  Quantification of vector copy numbers on sorted cells population by q-PCR
Replication competent lentivirus (RCL) | yearly from 3 years to 15 years (from 11 to 15 yearly time points, only in case of Advers Events of Special Interest)
  Presence of RCL
Change in medical conditions | yearly from 3 years to 10 years
  Weight and complete clinical exam
Key medical events related to WAS | yearly from 3 years to 10 years
  Eczema status, infections, bleeding symptoms, autoimmune manifestation
Hematological reconstitution | yearly from 3 years to 10 years
  CBC including platelets count and size
Reconstitution of cell mediated and humoral immunity | yearly from 3 years to 10 years (from 3 years to 5 years for PHA and candida )
  Immunophenotyping panel, whole blood lymphocytes proliferation assays, restoration of antibody production, humoral response to antigene

SECONDARY OUTCOMES:
Need for associated treatments | yearly from 3 years to 15 years
  Immunoglobulins, antibacterial, antifungal, antiviral drugs, transfusions
Representation of TCR families | yearly from 3 years to 5 years
  Representation of TCR families by PCR TREC (TCR excision circle) and TCR V beta panel
Bone marrow content | yearly from 3 years to 5 years (optional)
  Numbers and type of cells in bone marrow

CONTACTS AND LOCATIONS:
Locations (2):
- Hopital Necker - Enfants Malades, Paris, France
- UCL Institute of Child Health, London, United Kingdom

REFERENCES:
- [Derived] Magnani A, Semeraro M, Adam F, Booth C, Dupre L, Morris EC, Gabrion A, Roudaut C, Borgel D, Toubert A, Clave E, Abdo C, Gorochov G, Petermann R, Guiot M, Miyara M, Moshous D, Magrin E, Denis A, Suarez F, Lagresle C, Roche AM, Everett J, Trinquand A, Guisset M, Bayford JX, Hacein-Bey-Abina S, Kauskot A, Elfeky R, Rivat C, Abbas S, Gaspar HB, Macintyre E, Picard C, Bushman FD, Galy A, Fischer A, Six E, Thrasher AJ, Cavazzana M. Long-term safety and efficacy of lentiviral hematopoietic stem/progenitor cell gene therapy for Wiskott-Aldrich syndrome. Nat Med. 2022 Jan;28(1):71-80. doi: 10.1038/s41591-021-01641-x. Epub 2022 Jan 24. PMID 35075289